CLINICAL TRIAL: NCT00348985
Title: A Phase 1 Study of PXD101 in Combination With Bortezomib (PS-341) in Patients With Advanced Solid Tumors and Lymphoma
Brief Title: PXD101 and Bortezomib in Treating Patients With Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01052; COMIRB 05-0705; UCHSC-COMIRB-05-0705; UCHSC-05-0705; NCI-7281; CDR0000476293; U01CA099176 (NIH)
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Primary Central Nervous System Hodgkin Lymphoma; Primary Central Nervous System Non-Hodgkin Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — belinostat; Bortezomib

ARMS (1):
- PXD101 in Combination with Bortezomib (PS-341) (Experimental): Patients receive PXD101 IV over 30 minutes on days 1-5 and bortezomib IV on days 1, 4, 8, and 11 (2, 5, 8, and 11 during course 1).
  Interventions: Drug: belinostat; Drug: bortezomib; Other: pharmacological study

INTERVENTIONS:
Drug: belinostat
  Other Names: PXD101
Drug: bortezomib
  Other Names: LDP 341; MLN341; VELCADE
Other: pharmacological study
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of PXD101 and bortezomib in treating patients with advanced solid tumors or lymphomas. PXD101 and bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. PXD101 may also cause cancer cells to look more like normal cells, and to grow and spread more slowly. Giving PXD101 together with bortezomib may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Evaluate the safety profile and determine the maximum tolerated dose of PXD101 in combination with bortezomib in patients with advanced solid tumors or lymphomas.

II. Determine the pharmacokinetics of the combination of PXD101 and bortezomib in these patients.

III. Evaluate selected biomarkers of drug effect in these patients. IV. Evaluate the activity of this regimen, in terms of objective response rate, in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive PXD101 IV over 30 minutes on days 1-5 and bortezomib IV on days 1, 4, 8, and 11 (2, 5, 8, and 11 during course 1). Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-9 patients receive escalating doses of bortezomib and PXD101 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Blood is collected at baseline and periodically during course 1 of study treatment for pharmacokinetic studies.

After completion of study treatment, patients are followed periodically for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor or lymphoma that is refractory to standard therapy or for which no standard therapy exists
* No active, untreated, or symptomatic brain metastases

  * Patients with treated brain metastases are eligible provided metastasis are stable and the patient is off all steroids and anticonvulsants
* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN in the presence of liver metastases)
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to PXD101, bortezomib, boron, or mannitol
* No peripheral neuropathy > grade 1
* No uncontrolled intercurrent illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Psychiatric illness or social situation that would preclude study requirements
* No significant cardiovascular disease, including any of the following:

  * Myocardial infarction within the past 6 months
  * New York Heart Association class III-IV heart failure
  * Unstable angina pectoris
  * Uncontrolled hypertension
  * Condition requiring antiarrhythmic therapy
  * Ischemic or severe valvular heart disease
  * Acute ischemia or active conduction system abnormalities by ECG
* No marked baseline prolongation of QT/QTc interval (repeated demonstration of a QTc interval > 500 msec), long QT syndrome, or required use of concurrent medication during PXD101 administration that may cause torsade de pointes
* No severe medical or psychiatric problems of that would preclude study compliance
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, carmustine, or mitomycin C)
* At least 4 weeks since prior radiotherapy and recovered
* At least 2 weeks since prior palliative radiotherapy to sites involving < 35% of bone marrow reserve
* At least 4 weeks since prior investigational agents
* At least 2 weeks since prior valproic acid or any other histone deacetylase inhibitor
* No prior stem cell or bone marrow transplantation
* No concurrent radiotherapy or immunotherapy
* No concurrent hormonal therapy

  * Luteinizing hormone-releasing hormone agonists, selective estrogen receptor modulators, or aromatase inhibitors as chronic maintenance therapy allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of PXD101 in combination with bortezomib | Day 21
  Defined as the dose level below that which results in drug-related dose limiting toxicity (DLT) in >= 2 of 6 new patients.
Frequency and severity of treatment-related adverse events graded per NCI CTCAE version 3.0 | Day 21
Changes in biological markers (p21, cleaved PARP, IkB, p65 Rel A, p-AKT, p-ERK and apoptosis) from pre- to post-treatment | Baseline and day 21
Objective response rate | 4 weeks

SECONDARY OUTCOMES:
Pharmacokinetics of the combination of PXD101 with bortezomib | Baseline, end of infusion, then 15 minutes, 30 minutes, 1, 2, 4 and 6 hours from the end of infusion (days 1 and 2)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Eckhardt, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Colorado, United States